CLINICAL TRIAL: NCT01641510
Title: Phase 3 Study Comparing the Efficacy and Safety of Prasugrel and Clopidogrel in Acute Coronary Syndrome Patients With CYP2C19 Polymorphism Who Undergo Percutaneous Coronary Intervention.
Brief Title: PRAsugrel or clopIdogrel In Acute Coronary SyndromE With CYP2C19 GENEtic Variants
Acronym: PRAISE-GENE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Moo Hyun Kim, MD. Director, Regional Clinical Trial Center. Professor, Dept. of Cardiology Dong-A University Hospital, Dong-A University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRAISE-GENE
Record Dates: First submitted 2012-07-02; First posted 2012-07-16 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Acute Coronary Syndromes
Keywords: reduced-function CYP2C19 allele; high platelet reactivity; clopidogrel; prasugrel
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel (Experimental): Loading and maintenance dose of prasugrel
  Interventions: Drug: Prasugrel
- Clopidogrel (Active Comparator): Loading and maintenance dose of clopidogrel
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel — Loading with prasugrel 30 mg followed by daily administration of prasugrel 5 mg
  Other Names: Effient
  Arms: Prasugrel
Drug: Clopidogrel — Loading with clopidogrel 600 mg followed by daily administration of clopidogrel 75 mg
  Other Names: Plavix; Plavitor
  Arms: Clopidogrel

SUMMARY:
The investigators hypothesize that reduced loading dose of prasugrel followed by reduced maintenance dose of prasugrel in acute coronary syndrome patients with CYP2C19 polymorphism undergoing percutaneous coronary intervention might exhibit lower platelet reactivity 24 hours and 30 days later which is associated with major adverse cardiovascular events.

DETAILED DESCRIPTION:
Antiplatelet treatment is recommended worldwide for the secondary prevention and clopidogrel is an essential drug. But clopidogrel has limited value because of its pharmacodynamic interpatient variability and delayed onset time.

It is well known that patients who carry a common reduced-function CYP2C19 allele have a lower level of active metabolite of clopidogrel, diminished platelet inhibition, and furthermore, higher rate of major adverse cardiovascular events than noncarriers.

To achieve maximum plateau more rapidly and reduce the rate of high on-treatment platelet reactivity, higher loading dose of clopidogrel, up to 600 mg, is recommended. Although, however, the higher loading dose of clopidogrel, many patients still remain as non-responder.

Incidence of patients with clopidogrel resistance, especially CYP2C19*2 and *3, which encounter loss function, is higher in Eastern Asian peoples than Western peoples. Some studies report incidence rate of clopidogrel resistance in Eastern Asian peoples up to 99%.

However, the metabolism is not influenced by the presence of CYP2C19 genetic variation and prasugrel shows potent platelet inhibition. Although prasugrel exhibit potent platelet inhibition, recent reports describe the possible over inhibition of platelet especially in the East Asian people.

The investigators are going to compare the efficacy and safety of loading dose of prasugrel 30 mg which is lower than conventional loading dose followed by 5 mg/day which is also lower than conventional maintenance dose for 30 days and loading dose of clopidogrel 600 mg followed by 75 mg/day for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome
* Patients planned to undergo percutaneous transluminal coronary angioplasty
* Patients who agreed to the experimental plan which was permitted by IRB

Exclusion Criteria:

* Low body weight (< 50kg)
* History of stroke or transient ischemic attack
* History of upper gastrointestinal bleeding in recent 6 months
* Renal dysfunction defined by serum creatinine > 2.5 mg/dl
* Severe hepatic dysfunction defined by Child-Pugh criteria B or C
* Bleeding tendency
* Anticoagulation treatment including warfarin
* Thrombocytopenia defined by platelet < 100,000/ml
* Anemia defined by hemoglobin < 10 g/dl
* Contraindication for antiplatelet treatment or anticoagulation treatment
* History of administer glycoprotein IIb/IIIa inhibitor in recent 24hrs or planned to

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-10; Primary Completion 2018-10 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
HPR 1 day | 24 hours after PCI
  High platelet reactivity unit defined as platelet reactivity of 242u or more using VerifyNow method at 24 hours after PCI

SECONDARY OUTCOMES:
MACE | 30 days
  Major adverse cardiovascular events consist of cardiac death, myocardial infarction, stroke, stent thrombosis, cardiac enzyme (CRP, CK-MB, Troponin-I)
Bleeding | 30 days
  Major, minor or minimal bleeding defined by TIMI(thrombolysis in myocardial infarction) bleeding criteria
HPRs | 4 hours after PCI, 30 days after PCI
  High platelet reactivity unit defined as platelet reactivity of 240u or more using VerifyNow method at 4 hours and 30 days after PCI
HPR by VASP at 24 hours | 24 hours from PCI
  HPR defined by VASP at 24 hours after PCI
HPR by VASP at 30 days | 30 days from PCI
  HPR by VASP at 30 days from PCI

CONTACTS AND LOCATIONS:
Overall Officials: Moo Hyun Kim, MD, Principal Investigator — Director, Regional Clinical Trial Center
Locations (1):
- DongA University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided